CLINICAL TRIAL: NCT03902704
Title: Safety and Efficacy Assessment of a New Tracheal Intubation Device Cleverscope. Success Rate of Cleverscope in Patients With Suspected Difficult Airway.
Brief Title: Safety and Efficacy of Cleverscope. A New Medical Device for Tracheal Intubation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital General Universitario de Valencia (Other)
Collaborators: FIPSE (Unknown)
Responsible Party: Principal Investigator, Lucas Rovira, Principal Investigator, Hospital General Universitario de Valencia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Rov-Clever-2017
Record Dates: First submitted 2019-03-31; First posted 2019-04-04 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-05

CONDITIONS: Anesthesia Intubation Complication; Difficult Intubation
Keywords: videolaryngoscopy; tracheal intubation
MeSH Terms: interventions — Laryngoscopes

STUDY DESIGN:
Intervention Model Description: part 1 its single group of participants(50 patients without difficult airways predictors). this group receives direct laringoscopy with common laryngoscope (L) during the initial phase of the trial, followed by videolaryngoscope (VL) Cleverscope (used for intubation) during a later phase.
  part 2 of the study its two-by-two cross-over assignment involves two groups of participants(84 patients with difficult airways predictors). One group receives VL with C-MAC during the initial phase of the trial, followed by Cleverscope for intubation during a later phase. The other group receives VL with Cleverscope during the initial phase, followed by C-MAC VL used for intubation. So during the part 2 trial, participants "cross over" to the other videolaringoscopy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cleverscope (Experimental): Cleverscope is a new videolaryngoscope used for tracheal intubation. in this group we use this device to intubate participants.
  Interventions: Device: Cleverscope
- Laryngoscope / Videolaryngoscope C-MAC® Storz (Active Comparator): in this group we use a standart comercial device for intubation (laryngoscope or C-MAC) to intubate participants
  Interventions: Device: Laryngoscope / Videolaryngoscope C-MAC® Storz

INTERVENTIONS:
Device: Cleverscope — the device is used in patients without difficult airways predictors
  Arms: Cleverscope
Device: Laryngoscope / Videolaryngoscope C-MAC® Storz — the device is used in patients with difficult airways predictors
  Arms: Laryngoscope / Videolaryngoscope C-MAC® Storz

SUMMARY:
Cleverscope is a new medical device that transform a laryngoscope into a videolaryngoscope. previous its commercialization we evaluate its safety and efficacy.

DETAILED DESCRIPTION:
the investigators develope two part study. part I: the investigators collect data of 50 patients prospectively programed for general anesthesia and tracheal intubation without predictors of difficult airways. this patients were intubated with cleverscope, the investigators register best cormack-lehane (glottic vision) obtained with Cleverscope and best cormack obtained with direct laryngoscopy. the investigators register intubation succes rate and any complications during its use and after extubation.

part II: after confirm safety and efficacy in patients without difficult airways (part I) the investigators use Cleverscope for the same pourpose on difficult airways patients. collecting same data . the investigators compare cormack-lehane in this patients with Cleverscope and commercial Videolaryngoscope C-MAC.

ELIGIBILITY:
Inclusion Criteria:

* part 1: Scheduled Patients for any kind of surgery with general anesthesia with tracheal intubation without predictors of difficult intubation :

  1. Arne Test < 10
  2. cervical circunference / tyromental distance < 4.
* part 2: Scheduled Patients for any kind of surgery with general anesthesia with tracheal intubation with predictors of difficult intubation :

  1. Arne Test > 10
  2. cervical circunference / tyromental distance > 4.

Exclusion Criteria:

* no mouth openning >2cm
* required use of awake fiberscope por tracheal intubation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Cormack-Lehane Glotic visualization scale (I(complete view, easy to intubate)-IV(no view, imposible to intubate) | intraoperative
  degree of glotis visualization

SECONDARY OUTCOMES:
First attempt intubation success rate | intraoperative
  the rate of traqueal tube pass through vocal cords at first attemps.
overall success intubation rate with same device | intraoperative
  it could include more attempts
time to success | intraoperative
  time wasted from device inserted into mouth to inflate tracheal tube
complications rate | intraoperative
  register complications during intubation or due device usage. like hemorrage, mucosal laceration,

CONTACTS AND LOCATIONS:
Locations (1):
- Lucas Rovira, La Pobla de Vallbona, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No